CLINICAL TRIAL: NCT07231484
Title: Effects of Grape Consumption on Immune and Gut Health in the Setting of Obesity
Brief Title: Effects of Grape Consumption on the Immune-Gut Axis in Obesity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Principal Investigator, Jaapna Dhillon, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2128808
Record Dates: First submitted 2025-09-15; First posted 2025-11-17 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Obesity &Amp; Overweight
Keywords: Obesity; Immunity; Microbiome; Gut; Grape; Stress
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1: Grape then Placebo (Experimental): Whole freeze-dried grape powder for 4 weeks, 4-week washout, then isocaloric placebo powder for 4 weeks.
  Interventions: Other: Freeze-dried grape powder; Other: Placebo powder
- Sequence 2: Placebo then Grape (Experimental): Isocaloric placebo powder for 4 weeks, 4-week washout, then whole freeze-dried grape powder for 4 weeks.
  Interventions: Other: Freeze-dried grape powder; Other: Placebo powder

INTERVENTIONS:
Other: Freeze-dried grape powder — 48 g/day oral consumption during the 4-week active period.
Other: Placebo powder — Isocaloric placebo matched to grape powder; oral consumption during the 4-week active period.

SUMMARY:
This study is investigating the benefits of whole freeze-dried grape powder consumption on the immune-gut axis in adults with obesity.

DETAILED DESCRIPTION:
The study is a 12-wk randomized, controlled, crossover trial. Participants will be randomized to one of two intervention sequences, either consuming 48g/day of whole freeze-dried grape powder followed by an isocaloric placebo powder or consuming the placebo powder followed by the whole freeze-dried grape powder. Active intervention phases will be 4 weeks in duration followed by a 4-week washout period between treatments.

ELIGIBILITY:
Inclusion Criteria:

* Age: 30-45 years
* Obesity with BMI of 30-45 kg/m2
* Willingness to consume study foods
* Consistent diet and activity patterns for 4 weeks
* Weight stable (<5kg change over last 3 months)
* Non-smoker > 1 year or more
* Not currently consuming an extremely healthy diet

Exclusion Criteria:

* Study food allergies
* Regular consumption of grapes or grape-derived products
* Gastrointestinal disease and/or bariatric surgery
* Uncontrolled hypertension and blood pressure >180/110
* Diabetes
* Clinical Depression
* Illicit drug use
* History of alcohol or drug abuse
* Recent use of medications that affect immune function (e.g., corticosteroids)
* Recent consumption of antibiotics, prebiotics, probiotics, symbiotics, or dietary supplements containing fiber or phytochemicals
* Pregnant or lactating individuals
* HIV positivity
* Recent start of medications that affect metabolism or appetite
* Drug therapy for coronary artery disease, peripheral artery disease, congestive heart failure, or dyslipidemia

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Gut microbial diversity | Baseline, Week 4, Week 8, Week 12
  Assessed via 16s rRNA sequencing
LPS-binding protein concentration | Baseline, Week 4, Week 8, Week 12
  Intestinal permeability marker
Cytokine concentrations following PBMC stimulation | Baseline, Week 4, Week 12
  IL-6, IL-10
Perceived stress score | Baseline, Week 4, Week 8, Week 12
  Assessed using validated Cohen's Perceived Stress Scale. Scores range from 0-56 with higher scores indicating greater stress perceptions.

SECONDARY OUTCOMES:
Gut microbiome abundance | Baseline, Week 4, Week 8, Week 12
  Assessed via 16s rRNA sequencing
Inflammatory Markers | Baseline, Week 4, Week 8, Week 12
  IL-6, IL-10, TNF-alpha, IFN-gamma
Body mass | Baseline, Week 4, Week 8, Week 12
  Measured in kg
Body composition | Baseline, Week 4, Week 8, Week 12
  Fat mass and fat-free mass
Anthropometrics | Baseline, Week 4, Week 8, Week 12
  Waist circumference, hip circumference, thigh circumference
Glucoregulation | Baseline, Week 4, Week 8, Week 12
  Fasting glucose concentrations
Insulinemic biomarker concentrations | Baseline, Week 4, Week 8, Week 12
  Insulin concentrations
Lipid profile | Baseline, Week 4, Week 8, Week 12
  LDL, HDL, triglycerides, total cholesterol
Blood pressure | Baseline, Week 4, Week 8, Week 12
  Diastolic and systolic blood pressure
Dietary intake using 24-hour recalls | Every week
  24-hour diet recall using Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA-24).
Physical activity | Baseline, Week 4, Week 8, Week 12
  Activity assessment using Actigraphs
Sleep indices from Actigraphs | Baseline, Week 4, Week 8, Week 12
  Assessed using Actigraphs
24-hour appetite ratings | Baseline, Week 4, Week 8, Week 12
  24-hour appetite ratings assessed using Visual Analog Scale. For each question scores range from 0-100 with higher scores indicating "extremely" and lower scores indicating "not at all."
Palatability rating of foods | Every week
  Hedonic general labelled magnitude scale (gLMS). Scores range from 0 to 100.
Acceptance rating of foods | Every week
  9-point food action rating scale (1-9) with higher scores indicating a higher food rating.
Dietary Intake over past month | Baseline, Week 4, Week 8, Week 12
  Assessed using Food Frequency Questionnaires
IPAQ Score | Baseline, Week 4, Week 8, Week 12
  Measured using the International Physical Activity Questionnaire (IPAQ). Activity levels categorized as high, moderate, or low based on IPAQ scoring procedure.
Sleep indices from sleep diary | Baseline, Week 4, Week 8, Week 12
  Assessed using sleep diary

OTHER OUTCOMES:
Memory indices | Baseline, Week 4, Week 8, Week 12
  Assessed using memory tests
Attention indices | Baseline, Week 4, Week 8, Week 12
  Assessed using d2 test of attention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported here after deidentification (ie; text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Immediately following publication. No end date.
Access Criteria: Data will be deposited in online repositories